CLINICAL TRIAL: NCT03135964
Title: The Study of Wound Dressings for Portable Negative Pressure Wound Therapy
Brief Title: The Study of Wound Dressings for Portable NPWT
Acronym: NPWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tainan Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990903
Record Dates: First submitted 2015-11-04; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pressure Ulcer; Diabetic Foot Ulcer
Keywords: NPWT; foam; gauze
MeSH Terms: conditions — Pressure Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- foam (Active Comparator): PU foam dressing from KCI
  Interventions: Device: filler dressing of NPWT
- gauze (Active Comparator): Polyhexamethylene biguamide (PHMB) impregnated gauze (Kerlix AMD, Covidien)
  Interventions: Device: filler dressing of NPWT

INTERVENTIONS:
Device: filler dressing of NPWT — a dressing or filler material is used to fit to the contours of a wound (which is covered with a non-adherent dressing film) .
  Other Names: KCI PU foam dressing; Kerlix AMD gauze

SUMMARY:
Introduction Negative pressure wound therapy (NPWT), also known as topical negative pressure, has become a popular therapy for the treatment of many acute and chronic wounds. In many randomized controlled trials(RCTs), NPWT also has benefit in diabetic foot ulcer and pressure ulcer. However, most studies used commercial VAC device in combined with polyurethane (PU) foam. It is not yet clear where NPWT combined with gauze as wound filler is as effective as the PU foam. This RCT evaluated the efficacy of the gauze and PU foam, two kinds of fillers routinely used in negative pressure wound therapy, on the healing of the diabetic lower-extremity ulcers and the pressure ulcer.

Methods From 2010/1 to 2015/01, the in-patient persons with difficult to heal diabetic ulcer or Grade 4 pressure ulcer were enrolled. These patients were divided into two groups randomly. The letter of consent was signed by the patient or patient's family. After debridement of the infective wound, the wound of experimental group was packed with a moistened Polyhexamethylene biguamide (PHMB) impregnated gauze (Kerlix AMD, Covidien). A noncollapsible drainage tube (Blake drain, Ethicon) was applied to the wound, and then sealed with 3M Tegaderm Film. The system was connected to a 1-bottle water-seal chest drainage system and to standard wall suction at 125 mmHg negative pressure. The dressing was changed at 72- to 96-hour intervals (twice a week) for a period of 3 weeks. To the control group, the PU foam dressing from KCI was packed and sealed to the wound with the same continuous wall suction at -125mmHg. Investigators observed and recorded the ulcer area twice a week on each time of changing dressing in the following 3 weeks. The percentage of wound area reduction(PWAR) was used as a predictor of wound healing. The repeated measuring data were analyzed using linear mixed mode with SPSS statistical software. This clinical study was approved and monitored by Institutional Review Board of Show Chwan Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* in-patient persons with the pressure ulcer or diabetic ulcer

Exclusion Criteria:

* Patient who has uncontrolled medical condition, such as sepsis, cellulitis
* Patient with diabetic ulcer who has severe PAOD untreated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The reduction rate of pressure ulcer size | up to 3weeks

SECONDARY OUTCOMES:
The reduction rate of diabetic foot ulcer size | up to 3weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chin Yu, Master, Study Director — Tainan Municipal Hospital
Locations (1):
- Tainan Municipal Hospital, Tainan, Taiwan